CLINICAL TRIAL: NCT05796596
Title: Effectiveness of a Virtual Reality Game for Pediatric Pain and Anxiety Management During Skin Prick Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV-child-pain
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acute Pain
Keywords: Children; Anxiety; Pain; Skin Prick Testing
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned to one of three conditions: VR distraction group, book distraction control group, and no distraction group. Random assignments were generated with a random numbers table before recruitment by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (VR) distraction (Experimental): Distraction intervention using a virtual environment
  Interventions: Behavioral: Experimental: Virtual Reality (VR) distraction
- Distraction by the book (Active Comparator): Distraction intervention using a book visualization
  Interventions: Behavioral: Active Comparator: Distraction by the book
- Usual care (No Intervention): Control group receiving usual care and no distraction.

INTERVENTIONS:
Behavioral: Experimental: Virtual Reality (VR) distraction — Children in the VR distraction group will begin interacting with the virtual environment (VE) 2 minutes prior to the skin prick test and will continue playing throughout. The VR environment is a game in which the child draw a 360 degree image.
  Arms: Virtual Reality (VR) distraction
Behavioral: Active Comparator: Distraction by the book — In the book distraction group, the child will be invited to find and count animals in various landscapes. The book will be given 2 minutes prior to the skin prick test and continued reading throughout.
  Arms: Distraction by the book

SUMMARY:
This study investigated the effectiveness of virtual reality (VR) distraction, compared to book distraction and no distraction, in reducing pain and anxiety during a medical procedure in a pediatric population: the skin prick test. Although this test has many advantages and is considered to be minimally invasive, it causes anxiety and painful discomfort in children. This study concerns children aged 4 to 7 years consulting for an allergic test. Outcome measures include pain score, level of anxiety, VR measures, and satisfaction questionnaires.

DETAILED DESCRIPTION:
The use of skin prick tests is considered a gold standard in the evaluation of allergic reactions. These tests involve depositing a drop or small amount of the allergen on the skin and pricking the skin to let the allergen penetrate the epidermis. Although this test has many advantages and is considered to be minimally invasive, it causes anxiety and painful discomfort for children. Managing pain and anxiety during skin prick testing is essential to prevent long-term adverse effects, especially in the case of future needle-stick interventions. To our knowledge, the studies investigating distraction methods effect on reducing anxiety and pain during skin prick tests in childrenremain limited. No study has yet investigated the value of VR as a distraction tool in this field.

We postulate a greater decrease in child pain and child and parent anxiety in the RV and book conditions compared to the control group. We also postulate a larger effect for the RV group compared to the book group. In the VR group, we postulate the absence of an increase in post-immersion cybersickness symptoms. In last, we postulated a good satisfaction to distractions proposed, with a best score for RV distraction.

ELIGIBILITY:
Inclusion Criteria:

* speaking French regularly,
* requiring a skin prick test

Exclusion Criteria:

* have an epilepsy disorder
* have blindness

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Child's perceived pain | T2 (right after the skin prick testing).
  Child's perceived pain during prick test. Measured with Face Pain Scale - Revised (FPS-R) that is a self-report measure of pain intensity developed for children. Scores range from 0 (not bad at all) to 10 (very bad). The higher the score, the greater the pain.
Child's behavioral pain assessment | During the skin prick testing.
  Child's behavioral pain assessment during skin prick testing. Measured with Face Legs Activity Cry Consolability (FLACC) that is behavioral pain assessment scale used for nonverbal or preverbal patients who are unable to self-report their level of pain. Scores range from 0 to 10. The higher the score, the greater the pain.
Change in child's state anxiety | T1 (before the skin prick testing), T2 (right after the skin prick testing).
  Child skin prick testing anxiety. Measured with Glasses Fear Scale (GFQ; heteroevaluation and completed by the parent). Scores range from 0 (no fear) to 5 (intense fear). The higher the score, the greater the fear.
Change in parent's state anxiety | T1 (before the skin prick testing), T2 (right after the skin prick testing).
  Parent skin prick testing anxiety. Measured with Glasses Fear Scale (GFQ). Scores range from 0 (no fear) to 5 (intense fear). The higher the score, the greater the fear.
Change in simulator sickness | T1 (before the skin prick testing for RV group only), T2 (right after the skin prick testing for RV group only).
  Measured with Simulator Sickness Questionnaire (SSQ) that is an instrument which is used to measure the extent to which children feel simulator sickness due to their immersion in VR (e.g., nausea, eye fatigue, dizziness, etc.).
Child satisfaction questionnaire | T2 (right after the skin prick testing for RV and Book groups only).
  Satisfaction questionnaire is a visual analogue scale to measure the degree of child satisfaction related to the distraction used during the skin prick testing. Scores range from 0 (very dissatisfied) to 100 (very satisfied).
Parent satisfaction questionnaire | T2 (right after the skin prick testing for RV and Book groups only).
  Satisfaction questionnaire is a visual analogue scale to measure the degree of parent satisfaction related to the distraction used during the skin prick testing. Scores range from 0 (very dissatisfied) to 100 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Céline Stassart, PhD, Principal Investigator — University of Liege
Locations (1):
- Clinique CHC MontLégia, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No